CLINICAL TRIAL: NCT06582563
Title: Study for Evaluation of Clinical Ranges of Whole Blood Clotting Times
Brief Title: Evaluation of Clinical Ranges of Whole Blood Clotting Times of Patients on Anticoagulants
Status: Not yet recruiting | Type: Observational
Sponsor: Perosphere Technologies Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-01-02-002
Record Dates: First submitted 2024-08-21; First posted 2024-09-03 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Blood Coagulation Disorder
MeSH Terms: conditions — Blood Coagulation Disorders | interventions — Whole Blood Coagulation Time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Whole Blood Clotting Time — Comparator

SUMMARY:
Whole blood clotting time measurements are to collect the clotting time ranges for DOAC-anticoagulated patients and assess their correlation with plasma drug levels (via anti-FXa assay).

DETAILED DESCRIPTION:
Primary objectives of the planned whole blood clotting time measurements are to collect the clotting time ranges for DOAC-anticoagulated patients and assess their correlation with plasma drug levels (via anti-FXa assay).

ELIGIBILITY:
Inclusion Criteria:

* In general, study participants must:

  1. Be informed of the nature of the study and provide written informed consent before any study-specific procedures are performed.
  2. Be 18- to 80-years-of-age, inclusive, at time of consent.
  3. Have suitable venous access for at least a single venipuncture.
  4. Eligible patients on anticoagulants must have taken their prescribed anticoagulant regularly at least for one month prior to study participation for inclusion

Exclusion Criteria:

* Eligible patients on anticoagulants must not:

  1. Other than the condition for which a DOAC was prescribed , have a personal or family history of clotting disorder or hematologic abnormality, such as excessive bleeding, joint hematoma, thrombovascular disease, thrombocytopenia, or any chronic condition requiring treatment with transfusions.
  2. Have a BMI> 40 or weight > 120kg.
  3. Suffer from renal or hepatic insufficiency.
  4. Suffer from any pathology that would contra-indicate in general DOAC medication.
  5. Have a history of unexplained syncope.
  6. Have a history within 6 months prior to Screening of peptic ulcer or gastrointestinal bleeding (including hematemesis, melena, or rectal bleeding).
  7. Consume more than 5 cigarettes per day.
  8. If female, have a history of excessive or dysfunctional uterine bleeding (unless the subject had a subsequent hysterectomy).
  9. If female is pregnant, breastfeeding, or planning to become pregnant during study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with rivaroxaban, apixaban, or edoxaban between the ages of 18 and 80 years old. A sufficient number (12 or above) of the patients are above 70 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Clotting times of whole blood samples, measured on Perosphere Technologies' PoC Coagulometer devices | Immediate
  Whole Blood Clotting Time

SECONDARY OUTCOMES:
Drug concentrations in collected blood samples as measured through anti-factor Xa (anti-Xa) assay | Immediate
  Drug concentration measurements

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven Hospital, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided